CLINICAL TRIAL: NCT00880009
Title: A PHASE 2, RANDOMIZED, OPEN-LABEL STUDY OF BOSUTINIB ADMINISTERED IN COMBINATION WITH LETROZOLE VS. LETROZOLE ALONE AS FIRST LINE THERAPY IN POST-MENOPAUSAL WOMEN WITH LOCALLY ADVANCED OR METASTATIC ER+/PR+/HER2- BREAST CANCER.
Brief Title: Study Evaluating Bosutinib-Letrozole Combination Versus Letrozole Alone In Post Menopausal Women With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3160A6-2207; B1871010 (Other: Alias Study Number); 2008-006252-21 (EudraCT Number)
Record Dates: First submitted 2009-04-08; First posted 2009-04-13 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — bosutinib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Combination of Bosutinib and Letrozole
  Interventions: Drug: Bosutinib; Drug: Letrozole
- 2 (Active Comparator): Letrozole
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Bosutinib — 400mg (4x100)mg tablets once daily during the active phase of treatment until Disease Progression, unacceptable toxicity or withdraw of consents occurs
  Arms: 1
Drug: Letrozole — 2.5 mg - one tablet per day- once daily during the active phase of treatment until Disease Progression, unacceptable toxicity or withdraw of consents occurs
  Arms: 1
Drug: Letrozole — 2.5 mg - one tablet per day- once daily during the active phase of treatment until Disease Progression, unacceptable toxicity or withdraw of consents occurs
  Arms: 2

SUMMARY:
This is a phase 2 study of bosutinib administered in combination with letrozole versus letrozole alone in post-menopausal women with breast cancer. This is a 2-part study. Subjects in part 1 will receive bosutinib and letrozole daily, and will be closely monitored for 28 days. The second part will proceed with subjects receiving a dose that is determined to be safe based on the safety evaluation of the first part. Eligible subjects will be randomly assigned to receive either bosutinib daily combined with daily letrozole, or daily letrozole alone for a specified period of time. Subjects will be followed up for survival after study drug discontinuation.

DETAILED DESCRIPTION:
This study was terminated on 19 April 2009 due to unfavorable risk benefit ratio of Bosutinib in combination with Letrozole including one confirmed Hy's law case. 37.5% of patients had treatment related liver events with the majority of severe events resulting in permanent study treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Surgically sterile or post-menopausal women.
* Confirmed pathologic diagnosis of breast cancer.
* Locally advanced or metastatic, or loco-regional recurrent breast cancer not amenable to curative treatment with surgery or radiotherapy.
* Documented ER+ and/or PgR+ and erbB2- tumor based on most recently analyzed biopsy, as documented by a local laboratory.
* At least 1 radiologically measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

* Prior letrozole (except in adjuvant setting), prior bosutinib, or any other prior Src inhibitor.
* Prior endocrine treatment for locally advanced or metastatic breast cancer (up to one prior adjuvant Aromatase Inhibitor (AI) agent/regimen is permitted).
* More than 1 prior chemotherapy regimen in locally advanced or metastatic breast cancer.
* Adjuvant endocrine therapy <=12 months prior to day 1 of treatment.
* Disease refractory (ie, Progressive disease (PD) within 6 months from initiation of therapy) to previous adjuvant antiestrogen therapy.
* Bone or skin as the only site of disease.
* Extensive visceral disease or active Central Nervous System (CNS) disease.
* Any other cancer within 5 years of screening with the exception of ER+ contralateral breast carcinoma, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin.
* Major surgery or radiotherapy within 14 days of treatment day.
* Inadequate hepatic/renal/bone marrow function.
* History of clinically significant or uncontrolled cardiac disease.
* Serious concurrent illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2009-07-30 (Actual); Primary Completion 2010-05-31 (Actual); Study Completion 2010-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (5):
  - American Institute of Research, Whittier, California
  - Joliet Oncology Hematology Associates, Joliet, Illinois
  - Oncology Specialists SC, Niles, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
- AZ Sint-Augustinus, Wilrijk, Belgium
- Cancer Hospital, Academy of Med Science and Peking Union Med, Beijing, Beijing Municipality, China
- UNIMED Medical Institute, Hong Kong, Hong Kong
- Orszagos Onkologiai Intezet "B" Belgyogyaszati osztaly, Budapest, Hungary
- Centrum Medyczne Ostrobramska Niepubliczny Zaklad Opieki Zdr, Warsaw, Poland
- Johns Hopkins Singapore International Medical Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Moy B, Neven P, Lebrun F, Bellet M, Xu B, Sarosiek T, Chow L, Goss P, Zacharchuk C, Leip E, Turnbull K, Bardy-Bouxin N, Duvillie L, Lang I. Bosutinib in combination with the aromatase inhibitor letrozole: a phase II trial in postmenopausal women evaluating first-line endocrine therapy in locally advanced or metastatic hormone receptor-positive/HER2-negative breast cancer. Oncologist. 2014 Apr;19(4):348-9. doi: 10.1634/theoncologist.2014-0021. Epub 2014 Mar 27. PMID 24674874
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A6-2207&StudyName=Study%20Evaluating%20Bosutinib-Letrozole%20Combination%20Versus%20Letrozole%20Alone%20In%20Post%20Menopausal%20Women%20With%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was pre-maturely terminated after part 1 (safety lead-in phase) of the study and hence, the planned treatments of part 2, bosutinib + letrozole (Part 2) and letrozole (Part 2), were not administered.
Groups:
- Bosutinib + Letrozole (Part 1): Four bosutinib 100 milligram (mg) tablets, equivalent to 400 mg bosutinib along with letrozole 2.5 mg tablet orally once daily until disease progression, unacceptable toxicity or withdrawal of consent occurred.
Period: Overall Study
Arm/Group | Bosutinib + Letrozole (Part 1)
Started | 16
Completed | 0
Not Completed | 16
Not completed — Study terminated by sponsor | 14
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bosutinib + Letrozole (Part 1)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Based on Independent Radiologist
Description: Time in weeks from date of randomization to first documentation of objective tumor progression or death due to any cause. PFS: calculated as (first event date minus the date of randomization plus 1) divided by 7. Tumor progression: determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death"). PFS assessed by independent radiologist was to be reported.
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: Data were not analyzed because the study was prematurely terminated due to unfavorable risk benefit ratio of the study treatment.
Groups:
- Bosutinib + Letrozole (Part 2): Four bosutinib 100 mg tablets, equivalent to 400 mg bosutinib along with letrozole 2.5 mg tablet orally once daily until disease progression, unacceptable toxicity or withdrawal of consent occurred.
- Letrozole (Part 2): Letrozole 2.5 mg tablet orally once daily until disease progression, unacceptable toxicity or withdrawal of consent occurred.
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Part 1 Baseline up to 28 days after the last dose
Population: Safety population included all participants who receive at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib + Letrozole (Part 1)
Number analyzed (Participants) | 16
percentage of participants
  AEs | 100
  SAEs | 31.3

3. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator
Description: Time in weeks from date of randomization to first documentation of objective tumor progression or death due to any cause. PFS: calculated as (first event date minus the date of randomization plus 1) divided by 7. Tumor progression: determined from oncologic assessment data (where data meet the criteria for PD), or from AE data (where the outcome was "Death"). PFS assessed by investigator was to be reported.
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as greater than or equal to >=30 percent (%) decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from randomization to date of death due to any cause. OS was calculated as (the death date minus the date of randomization plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Part 2 Baseline until death or up to 36 months
Population: as for outcome 1
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 1
Groups:
- Bosutinib + Letrozole (Part 2): Four bosutinib 100 milligram (mg) tablets, equivalent to 400 mg bosutinib along with letrozole 2.5 mg tablet orally once daily until disease progression, unacceptable toxicity or withdrawal of consent occurred.
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B)
Description: FACT-B is used for assessment of health-related quality of life (QoL) in participants with breast cancer. It consists of 36 items, summarized to 5 subscales: physical (7 items), functional (7 items), social/family (7 items); all 3 ranged from 0 to 28, emotional (6 items) ranging from 0 to 24, and additional concerns on breast cancer subscale (9 items) ranging from 0 to 36; high subscale score represents a better QoL. All single-item measures ranges from 0='Not at all' to 4='Very much'. Total possible score ranged from 0 to 144. High scale score represents a better QoL.
Time Frame: Part 2 Baseline, Week 12, 24, 52, 2-6 weeks after the last dose
Population: as for outcome 1
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 hour (pre-dose) on Day 1; 2, 3, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 1
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 hour (pre-dose) on Day 1; 2, 3, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 1
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)]
Description: AUC (0-24)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24).
Time Frame: 0 hour (pre-dose) on Day 1; 2, 3, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 1
Arm/Group | Bosutinib + Letrozole (Part 2) | Letrozole (Part 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bosutinib + Letrozole (Part 1)
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib + Letrozole (Part 1) (N=16)
Myocardial ischaemia (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib + Letrozole (Part 1) (N=16)
Lymphopenia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 13
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 4
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 1
Blood creatinine (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Deep vein thrombosis (Vascular disorders) | 1
Hot flush (Vascular disorders) | 3
Hypertension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Results are not provided because the study was terminated prior to part 2 due to unfavorable risk benefit ratio of the study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.